CLINICAL TRIAL: NCT00571948
Title: Dortmund Intervention Trial for Optimization of Infant Nutrition
Brief Title: Modification in Complementary Food Composition to Improve the Status of Iron and Fatty Acids in Infants.
Acronym: DINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute of Child Nutrition, Dortmund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2XIKers
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Iron Status; Fatty Acid Status
Keywords: infant, complementary food, iron, meat, LC-PUFA, omega-3,; rapeseed oil, diet
MeSH Terms: interventions — Fatty Acids, Omega-3; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Babyfood with usual meat content and corn oil (Active Comparator): Infants in the control group received vegetable-potato-meat-meals as part of complementary food containing common amounts of meat and corn oil marketed in Germany.
  Interventions: Other: more meat and a vegetable oil rich in omega-3 fatty acids; Other: Babyfood with usual meat content and corn oil
- more meat and a vegetable oil rich in omega-3 fatty acids (Experimental): Infants in the intervention group received vegetable-potato-meat-meals as part of complementary food containing higher amounts of meat than the control group and rapeseed oil instead of corn oil.
  Interventions: Other: more meat and a vegetable oil rich in omega-3 fatty acids; Other: Babyfood with usual meat content and corn oil

INTERVENTIONS:
Other: more meat and a vegetable oil rich in omega-3 fatty acids — The vegetable-potato-meat-meal was given 5 to 7 times a week for at least during the seventh to tenth month.
  The intervention meals had more meat (about 13 % of weight) and rapeseed oil (rich in omega-3 fatty acids).
Other: Babyfood with usual meat content and corn oil — The active comparator (which is the control group) got babyfood with usual meat content (8%) and with corn oil, which is rich in omega 6 linoleic acid

SUMMARY:
The objective of this study is to determine the influence of an increase of meat in complementary food on iron status and the effect of an exchange of vegetable oil in the same food on the status of omega-3 fatty acids in infants in the second six months of life.

DETAILED DESCRIPTION:
Because of rapid growth in the first year of life, infants are at a high risk to develop iron deficiency (ID) or even iron deficiency anaemia (IDA). Iron metabolism in infancy seems to be immature and to be affected by developmental changes and is not yet fully understood. Therefore studies with both, detailed dietary intake and a full set of biomarkers to characterize iron status or the risk of IDA are welcome.

LC-PUFA, especially docosahexaenoic acid (DHA, n-3), are of important meaning in infants´ neural development because neural tissues have a unique pattern of FA. DHA is predominantly found in brain and retina. LC-PUFA can be either supplied preformed by diet or converted from their essential precursors the polyunsaturated fatty acids (PUFA) linoleic acid (LA, n-6) and α-linolenic acid (ALA, n-3) by the organism dependent on the ratio of n-6/n-3 FA in the diet.

In the case of iron as well as of PUFA and LC-PUFA very little is known about the nutritional supply and its effect on status in the second half of the first year of life. Therefore the objective of DINO is to examine the feasibility of increasing meat and of exchanging n-6 rich corn oil vs. n-3 rich rapeseed oil in common commercial menus and to examine the effects on iron status and on blood FA pattern respectively as primary outcome variables in a double-blinded randomized controlled intervention trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* a term healthy newborn infant (birth weight > 2500 g, gestational age > 37 weeks);
* inclusion during the first two months of life.
* German speaking mother;
* the intention of the mother to breast-feed the child and to feed study menus 5 to 7 times per week beginning in the fifth to seventh month of life.

Exclusion Criteria:

* preterm infants

Ages: 1 Week to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Kersting, PD Dr., Principal Investigator — Research Institute of Child Nutrition
Locations (1):
- Research Institute of Child Nutrition, Dortmund, Nord-Rhein-Westfalen, Germany

REFERENCES:
- [Result] Schwartz J, Dube K, Sichert-Hellert W, Kannenberg F, Kunz C, Kalhoff H, Kersting M. Modification of dietary polyunsaturated fatty acids via complementary food enhances n-3 long-chain polyunsaturated fatty acid synthesis in healthy infants: a double blinded randomised controlled trial. Arch Dis Child. 2009 Nov;94(11):876-82. doi: 10.1136/adc.2008.146027. Epub 2009 Feb 4. PMID 19193660
- [Result] Schwartz J, Dube K, Alexy U, Kalhoff H, Kersting M. PUFA and LC-PUFA intake during the first year of life: can dietary practice achieve a guideline diet? Eur J Clin Nutr. 2010 Feb;64(2):124-30. doi: 10.1038/ejcn.2009.123. Epub 2009 Nov 25. PMID 19935821
- [Result] Schwartz J, Drossard C, Dube K, Kannenberg F, Kunz C, Kalhoff H, Kersting M. Dietary intake and plasma concentrations of PUFA and LC-PUFA in breastfed and formula fed infants under real-life conditions. Eur J Nutr. 2010 Apr;49(3):189-95. doi: 10.1007/s00394-009-0067-1. Epub 2009 Oct 23. PMID 19851802
- [Result] Dube K, Schwartz J, Mueller MJ, Kalhoff H, Kersting M. Complementary food with low (8%) or high (12%) meat content as source of dietary iron: a double-blinded randomized controlled trial. Eur J Nutr. 2010 Feb;49(1):11-8. doi: 10.1007/s00394-009-0043-9. Epub 2009 Jul 19. PMID 19618230
- [Derived] Dube K, Schwartz J, Mueller MJ, Kalhoff H, Kersting M. Iron intake and iron status in breastfed infants during the first year of life. Clin Nutr. 2010 Dec;29(6):773-8. doi: 10.1016/j.clnu.2010.05.002. Epub 2010 Jun 2. PMID 20627488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers were first contacted in the hospital 1-3 days after delivery. Of 832 contacted families 132 agreed to participate in the study up to the baby's age of 8 weeks.
Pre-assignment Details: All of the 132 participants were randomly assigned to one of the two study groups.
Groups:
- Participants in the Control Group: Infants in the control group received vegetable-potato-meat-meals as part of complementary food containing common amounts of meat and corn oil marketed in Germany.
- Participants in the Intervention Group: Infants in the intervention group received vegetable-potato-meat-meals as part of complementary food containing higher amounts of meat than the control group and rapeseed oil instead of corn oil.
Period: Overall Study
Arm/Group | Participants in the Control Group | Participants in the Intervention Group
Started | 66 | 66
Completed | 55 (Excluded from analysis (n = 2) Reason: diet record for less than 75 % of days (n = 2)) | 52 (Excluded n = 3) Reasons: diet record < 75 % of days (n = 2); blood analysis failed (n= 1))
Not Completed | 11 | 14
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 3 | 3
Not completed — infant refused study meal | 3 | 4
Not completed — Parent were afraid of blood colection | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants in the Control Group | Participants in the Intervention Group | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Customized [Number; unit: Participants]
  <=2 months at beginning | 66 | 66 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 31 | 34 | 65
Region of Enrollment [Number; unit: participants]
  Germany | 66 | 66 | 132

OUTCOME MEASURES:

1. Primary Outcome: Sum of Omega-3 Fatty Acid Pattern in Plasma
Description: fatty acids were measured in the whole plasma (in mg). They were transformed into percent (%) per total fatty acids.
  Results are shown as percent (%) per total fatty acids before and after the intervention as median (percentile 25th;75th).
Time Frame: at the end of the tenth month of life
Measure: Median (Inter-Quartile Range); unit: percent of total fatty acids
Arm/Group | Participants in the Control Group | Participants in the Intervention Group
Number analyzed (Participants) | 55 | 52
percent of total fatty acids | 2.66 [2.33 to 2.87] | 3.02 [2.85 to 3.66]

2. Secondary Outcome: Dietary Intake; Anthropometric Measures: Body Weight, Body Lengths, Head Circumferences
Time Frame: dietary intake: from the beginning of the third month of life to the end of the tenth month; anthropometric measures: at the end of the fourth, seventh, tenth month
Reporting Status: Not Posted

3. Primary Outcome: Parameters of Iron Status in Blood
Time Frame: at the end of the fourth, seventh, tenth month of life
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Participants in the Control Group | Participants in the Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No